CLINICAL TRIAL: NCT01933386
Title: Evaluation of Benefit for Treatment of Single Sided Deafness (SSD) Between Two Bone Conduction Prosthetic Devices; Osseointegrated Implant Versus Maxilla Anchored Removable Oral Appliance ("SoundBite")
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sonitus Medical Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CLN008
Record Dates: First submitted 2013-08-28; First posted 2013-09-02 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-10

CONDITIONS: Single Sided Deafness
Keywords: Single Sided Deafness; SSD; Unilateral hearing loss
MeSH Terms: conditions — Hearing Loss, Unilateral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SoundBite (Other): SoundBite will be used for the first 30 days
  Interventions: Device: SoundBite
- Surgically Implanted BCD (Other): The subject's own surgically implanted bone conduction device will be used for the first 30 days.
  Interventions: Device: SoundBite

INTERVENTIONS:
Device: SoundBite — Non-surgical removable bone conduction device via the teeth.
  Other Names: The SoundBite Hearing System

SUMMARY:
The primary objective of this study is to compare the SoundBite™ Hearing System to surgically implanted BCD systems.

ELIGIBILITY:
Inclusion Criteria:

* Must be current users of a surgically implanted digitally programmable surgically implanted bone conduction device
* Must be >18, <80 years old
* Must be fluent in English, as determined by the PI
* Must have diagnosis of SSD, time since onset (≥3 months)
* Must have at least two contiguous molar or premolar teeth with no untreated tooth decay. Patients with tooth decay present are to first have restorations before being fitted for SoundBite
* Healthy attachment to those teeth with tooth pockets limited to no more than 5mm

Exclusion Criteria:

* Subjects with known hypersensitivity to any of the components including allergies to polymers.
* Subjects that are unable to use their hands such as quadriplegics or others that are unable to comply with the warnings in the product's labeling.
* Subjects with known or active secondary medical conditions associated with variable sensorineural hearing loss

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-02 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
APHAB Questionnaire | 30 days
  Comparison of the SoundBite™ System and surgically implanted bone conduction devices

SECONDARY OUTCOMES:
Single Sided Deafness Questionnaire | 30 days
  Comparison of the SoundBite™ System and surgically implanted BCD systems.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Syms, MD, Principal Investigator — Ear Medical Group
Locations (3):
- United States (3):
  - Arizona Ear Center, Phoenix, Arizona
  - Michigan Ear Institute, Novi, Michigan
  - Ear Medical Group, San Antonio, Texas

REFERENCES:
- See also: SoundBite Hearing System — http://soundbitehearing.com